CLINICAL TRIAL: NCT00540969
Title: A Phase III Randomized Trial of Cryoablation vs. Radiation for the Palliation of Painful Bone Metastases
Brief Title: Cryoablation or External-Beam Radiation Therapy in Treating Patients With Painful Bone Metastases
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N06C6; NCI-2009-00690 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000570788 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Kidney Cancer; Melanoma (Skin); Metastatic Cancer; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: bone metastases; pain; unspecified adult solid tumor, protocol specific; stage IV melanoma; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Neoplasm Metastasis; Pain; Carcinoma, Renal Cell | interventions — Cryosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (percutaneous cryoablation) (Experimental): Cryoprobes are inserted percutaneously under CT scan or ultrasound guidance, to the malignant soft tissue-bone interface. Patients undergo ablations using a freeze-thaw-freeze cycle lasting approximately 10-5-10 minutes, respectively.
  Interventions: Procedure: cryosurgery
- Arm II (external-beam radiotherapy) (Active Comparator): Patients undergo external-beam radiotherapy comprising either a single 8 Gy dose or 20 Gy/5 fractions administered over 1 week.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Procedure: cryosurgery — Patients undergo cryosurgery using guidance from CT scan or ultrasound
  Arms: Arm I (percutaneous cryoablation)
Radiation: radiation therapy — Patients undergo radiotherapy for 1 week
  Arms: Arm II (external-beam radiotherapy)

SUMMARY:
RATIONALE: Cryoablation kills cancer cells by freezing them. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. It is not yet known whether cryoablation is more effective than external-beam radiation therapy in treating painful bone metastases.

PURPOSE: This randomized phase III clinical trial is studying cryoablation to see how well it works compared with external-beam radiation therapy in treating patients with painful bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine pain relief in cancer patients with painful metastatic disease involving bone following treatment with cryoablation as compared to radiotherapy (RT).
* To compare the impact on quality-of-life following cryoablation or RT in patients with painful metastatic disease as measured using the validated Brief Pain Inventory (BPI) and Short Form (SF)-8.
* To determine change in analgesic use following therapy.
* To determine the frequency and severity of complications following treatment of painful metastases involving bone with either cryoablation or RT.

OUTLINE: This is a multicenter study. Patients are stratified according to size of the indexing lesion (≤ 5 cm vs > 5 cm), location of the target lesion (pelvis vs extremity vs vertebral body vs other), primary cancer type (melanoma or renal cell carcinoma vs other), and severity of pain (i.e., worst pain score in the last 24-hour period) (4-6 vs 7-10). Patients are randomized to 1 of 2 treatment arms.

* Arm I (percutaneous cryoablation): Cryoprobes are inserted percutaneously under CT scan or ultrasound guidance, to the malignant soft tissue-bone interface. Patients undergo ablations using a freeze-thaw-freeze cycle lasting approximately 10-5-10 minutes, respectively.
* Arm II (external-beam radiotherapy): Patients undergo external-beam radiotherapy comprising either a single 8 Gy dose or 20 Gy/5 fractions administered over 1 week.

Patients are contacted via phone on days 1 and 4 post treatment, weekly in weeks 1-4, every 2 weeks in weeks 6-24, and then every four weeks in weeks 28-36. Patients undergo pain and pain interference with daily life assessment at baseline and at these time points. Patients who elect to have repeated treatment (either radiotherapy or cryoablation) within the first 6 weeks after the initial treatment are removed from the study. Patients who fail to achieve a 2-point reduction in worst or average pain (in a 24-hour period) during weeks 6-20 after initial treatment and patients who report a return of pain (i.e., pain ≥ the worst pain in a 24-hour period reported at baseline) for 2 consecutive time points are offered the alternative treatment (radiotherapy or cryoablation, whichever the patient was not randomized to receive at initial treatment)*.

NOTE: *Patients who refuse to receive the alternative treatment are taken off study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed solid tumor metastasis with index lesion involving or abutting bone

  * Index lesion with bone destruction is predominantly osteolytic in nature as assessed on CT imaging
  * If the nature of the metastatic disease has been previously documented, the index lesion to be treated does not require further documentation (i.e., biopsy)
* One primary painful metastatic site

  * Additional less painful metastatic sites may be present
* Worst pain in the last 24 hours must be ≥ 4 on a 0-10 numeric scale
* Current analgesic therapies have failed OR the patient is experiencing intolerable side effects
* Tumor is appropriate for radiotherapy as determined by the participating radiation oncologist and accessible for cryoablation as determined by the participating radiologists upon review of ultrasound, CT scan, X-ray, or MRI examinations
* Have completed chemotherapy, hormonal therapy, or bisphosphonate therapy ≥ 4 weeks prior to registration OR have developed pain or have persistent pain while on a stable chemotherapy, hormonal therapy, or bisphosphonate therapy regimen for a period of ≥ 4 weeks

Exclusion criteria:

* Index lesion causing clinical or radiographic evidence of spinal cord or cauda equina compression/effacement
* Index lesion involves the skull

  * Treatment of other painful lesions in patients with skull lesions is not excluded
* Index lesion has evidence of a pathologic fracture or impending fracture in weight-bearing bones (e.g., vertebral body, periacetabular region, femur, or tibia) with > 50% loss of cortical bone

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 2 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* No concurrent medication known to interfere with platelet function or coagulation (e.g., aspirin, ibuprofen, clopidogrel, or warfarin) and such medications have been discontinued for an appropriate time period based on the drug half-life and known activity (e.g., aspirin for 7 days) for patients randomized to receive cryoablation only
* Low molecular weight heparin preparations must be discontinued 8 hours prior to cryoablation
* At least 2 weeks since prior cytotoxic chemotherapy (for patients randomized to receive cryoablation only)

Exclusion criteria:

* Has undergone prior cryoablation or radiotherapy of the index lesion
* Prior radiopharmaceutical therapy completed ≤ 4 weeks prior to registration
* Initiation of new chemotherapy ≤ 4 weeks prior to registration
* Concurrent surgery involving the treated lesion
* Anticipated treatment of the index lesion that would require ice-ball formation within 0.5 cm of the spinal cord, brain, other critical nerve structure, large abdominal vessel such as the aorta or IVC, bowel, or bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Callstrom, MD, PhD, Study Chair — Mayo Clinic
Locations (7):
- United States (7):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Percutaneous Cryoablation) | Arm II (External-beam Radiotherapy)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Percutaneous Cryoablation) | Arm II (External-beam Radiotherapy) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Pre- and Post-treatment Worst Pain in 24 Hours at Week 6 as Measured on the Numeric 0 to 10 Brief Pain Inventory (BPI) Scale
Time Frame: at week 6
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I (Percutaneous Cryoablation) | Arm II (External-beam Radiotherapy)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Average Difference in Pre- and Post-treatment Average Pain, Pain Relief, and Pain Interference Scores at Week 6 as Measured With the BPI
Time Frame: at week 6
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I (Percutaneous Cryoablation) | Arm II (External-beam Radiotherapy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Average Difference in Pre- and Post-treatment Physical (PCS-8) and Mental (MCS-8) Quality of Life at Week 6 as Measured by the 2 Subscales of the Short Form (SF)-8
Time Frame: at week 6
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I (Percutaneous Cryoablation) | Arm II (External-beam Radiotherapy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I (Percutaneous Cryoablation) | Arm II (External-beam Radiotherapy)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes